CLINICAL TRIAL: NCT01985672
Title: Vitamin D Deficiency and Pregnancy Rates in Women Undergoing Frozen Embryo Transfer. A Prospective Cohort Study
Brief Title: Vitamin D Deficiency and Pregnancy Rates in Women Undergoing Frozen Embryo Transfer
Status: Completed | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Nikolaos P. Polyzos, Principal Investigator, Universitair Ziekenhuis Brussel
Other Study IDs: 2013/181; B.U.N. 143201317807
Record Dates: First submitted 2013-11-10; First posted 2013-11-15 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Infertility
Keywords: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Vitamin D deficient patients: Serum 25-OH Vitamin D levels <20ng/L undergoing Frozen embryo transfer (vitamin D levels are measured on the day of embryo transfer)
  Interventions: Procedure: Frozen embryo transfer
- Vitamin D sufficient patients: Serum 25-OH Vitamin D levels >20ng/L undergoing Frozen embryo transfer (vitamin D levels are measured on the day of embryo transfer)
  Interventions: Procedure: Frozen embryo transfer

INTERVENTIONS:
Procedure: Frozen embryo transfer — Embryo transfer of frozen/thawed embryos after IVF/ICSI

SUMMARY:
Vitamin D receptors are present and differently expressed in murine endometrium and ovary throughout the estrous cycle , whereas knock-out experiments have shown that vitamin D receptor null mice experience uterine hypoplasia and impaired folliculogenesis.

Only few retrospective studies examining the role of vitamin D levels in infertile patients have been published up to date, whereas results are strongly contradictory, with some supporting that maternal vitamin D deficiency is associated with lower pregnancy rates and others demonstrating that vitamin D deficiency does not affect final reproductive outcome.

Finally, a recent retrospective study postulated that vitamin D deficiency may negatively affect pregnancy rates with an effect mediated through the endometrium, given that vitamin D deficiency was not correlated with ovarian stimulation characteristics or with markers of embryo quality in this study.

In order to examine a potential negative effect of vitamin D deficiency on pregnancy rates, mediated through the endometrium, the aim of the current study was to examine the impact of vitamin D levels on pregnancy rates only in an infertile population undergoing embryo transfer of frozen-thawed embryos.

ELIGIBILITY:
Inclusion Criteria:

* All women undergoing a frozen ET with 1 or 2 Day 5 (blastocyst stage) embryo
* Age 18-39

Exclusion Criteria:

* Women > or = 40 years old
* IVM ET
* Uterine abnormalities

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertile women undergoing a frozen ET with 1 or 2 Day 5 (blastocyst stage) embryo
Sampling Method: Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2013-08; Primary Completion 2014-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy | 4 weeks after embryo transfer
  The presence of intrauterine gestational sac at 7 weeks of gestation

SECONDARY OUTCOMES:
Biochemical pregnancy | 2 weeks after embryo transfer
  Positive pregnancy test 2 weeks after embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos P. Polyzos, MD PhD, Principal Investigator — Universitair Ziekenhuis Brussel; Arne Van de Vijver, MD, Principal Investigator — UZBrussel
Locations (1):
- Centre for Reproductive Medicine UZ Brussel, Brussels, Belgium

REFERENCES:
- [Background] Zarnani AH, Shahbazi M, Salek-Moghaddam A, Zareie M, Tavakoli M, Ghasemi J, Rezania S, Moravej A, Torkabadi E, Rabbani H, Jeddi-Tehrani M. Vitamin D3 receptor is expressed in the endometrium of cycling mice throughout the estrous cycle. Fertil Steril. 2010 May 15;93(8):2738-43. doi: 10.1016/j.fertnstert.2009.09.045. Epub 2009 Nov 6. PMID 19896660
- [Background] Yoshizawa T, Handa Y, Uematsu Y, Takeda S, Sekine K, Yoshihara Y, Kawakami T, Arioka K, Sato H, Uchiyama Y, Masushige S, Fukamizu A, Matsumoto T, Kato S. Mice lacking the vitamin D receptor exhibit impaired bone formation, uterine hypoplasia and growth retardation after weaning. Nat Genet. 1997 Aug;16(4):391-6. doi: 10.1038/ng0897-391. PMID 9241280
- [Background] Rudick B, Ingles S, Chung K, Stanczyk F, Paulson R, Bendikson K. Characterizing the influence of vitamin D levels on IVF outcomes. Hum Reprod. 2012 Nov;27(11):3321-7. doi: 10.1093/humrep/des280. Epub 2012 Aug 21. PMID 22914766
- [Background] Anifandis GM, Dafopoulos K, Messini CI, Chalvatzas N, Liakos N, Pournaras S, Messinis IE. Prognostic value of follicular fluid 25-OH vitamin D and glucose levels in the IVF outcome. Reprod Biol Endocrinol. 2010 Jul 28;8:91. doi: 10.1186/1477-7827-8-91. PMID 20667111
- [Background] Ozkan S, Jindal S, Greenseid K, Shu J, Zeitlian G, Hickmon C, Pal L. Replete vitamin D stores predict reproductive success following in vitro fertilization. Fertil Steril. 2010 Sep;94(4):1314-1319. doi: 10.1016/j.fertnstert.2009.05.019. Epub 2009 Jul 8. PMID 19589516
- [Background] Aleyasin A, Hosseini MA, Mahdavi A, Safdarian L, Fallahi P, Mohajeri MR, Abbasi M, Esfahani F. Predictive value of the level of vitamin D in follicular fluid on the outcome of assisted reproductive technology. Eur J Obstet Gynecol Reprod Biol. 2011 Nov;159(1):132-7. doi: 10.1016/j.ejogrb.2011.07.006. Epub 2011 Aug 10. PMID 21835540